CLINICAL TRIAL: NCT04546412
Title: Importance of the Microtubule Cytoskeleton in Oocyte Competence
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidade de Lisboa (Network)
Responsible Party: Sponsor
Other Study IDs: 1907-LIS-072-AP
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: ART
Keywords: Oocyte competence; Oocyte vitrification; Cryobiology; Microtubule cytoskeleton

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Consenting subjects will donate supernumerary mature oocytes for the study following exogenous ovarian stimulation. However, no genetic analyses will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fresh oocytes: Sibling oocytes not subjected to vitrification prior to assessment
- Vitrified-thawed oocytes: Sibling oocytes subjected to vitrification using the Cryotop® - Open System and thawing prior to assessment
  Interventions: Device: Vitrification and thawing

INTERVENTIONS:
Device: Vitrification and thawing — Vitrification using the Cryotop® - Open System followed by thawing
  Groups: Vitrified-thawed oocytes

SUMMARY:
This study will assess if there are microtubule cytoplasmic features specifically associated with oocyte vitrification.

DETAILED DESCRIPTION:
Successful fertilization is heavily dependent upon inherent qualities of the oocytes, and thus reliant upon the fidelity of oocyte maturation. Reduced oocyte developmental competence is one of the main reasons for the decreased potential of in-vitro-produced embryos. Approximately 8,6% to 15% of all infertility patients produce at least one meiotically incompetent oocyte. There are also extreme cases of women which generate oocytes with complete or predominant failure to complete meiosis. These oocytes arrest and do not complete meiosis in response to exogenous final maturation and ovulation triggering. The incidence of this is unknown, and given the complexity of the processes involved in oocyte maturation, it has been difficult to define the key events or morphological features underlying oocyte competence.

An increasing amount of evidence in the past years has suggested that the microtubule (MT) cytoskeleton may have an important role in providing the oocyte with competence potential. Oocyte maturation involves major rearrangements of the MT cytoskeleton. It is well known the importance of forming a proper microtubule meiotic spindle for chromosome segregation upon meiosis. Moreover, MTs seem to be important for the redistribution of different organelles upon maturation. However, the exact functional significance of this reorganization and how MTs influence competence through the repositioning of these organelles is largely unknown.

The main MT organizing center in eukaryotic cells is the centrosome. Indeed, centrosomes are essential for the formation of the mitotic MT bipolar spindle. Interestingly, in the vast majority of female eggs these structures are eliminated, and the meiotic spindle does not contain centrosomes. A recent study in the lab organism Drosophila melanogaster (fruit fly), showed that interrupting this elimination, forcing the maintenance of centrosomes up to meiosis, led to female infertility. Both meiosis and the first nuclear divisions upon fertilization showed abnormal MT spindles with abnormal chromosome congression. This shows that proper spaciotemporal MT organization is likely to have important implications on oocyte competence.

The long-term goal of this research group is to analyze the MT cytoskeleton of oocytes from women which, upon assisted reproductive technologies, generate a high percentage of arrested embryos. In order to do this, the MT features of already-available surplus and unused oocytes which are vitrified and available for research purposes will be compared. These oocytes were donated from cycles in which a low (<20% the fertilized embryos) and high (>20% the fertilized embryos) incidence of arrested embryos was seen. Previous studies have posited that oocyte vitrification and warming may expose the oocyte to a variety of physical and chemical processes which may impact on their structural and genomic integrity. Therefore, this initial feasibility pilot study will investigate potential structural consequences for the oocytes of the vitrification procedure used in house.

Thus, it will be assess whether the Cryotop® - Open System induces specific MT features which may be absent in fresh oocytes. In case that both fresh and vitrified oocytes (derived from the same patient - sibling oocytes study) show a similar MT cytoskeleton organization, a collection of cryopreserved oocytes donated for research purposes will be used in the planned future studies of this research group.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form dated and signed.
* Already consented to perform oocyte donation.
* Age ≥18 and <35 years old.
* AFC ≥20.
* BMI ≥18.5 Kg/m2 and <30 Kg/m2.
* Two ovaries present.
* No current pregnancy-wish.

Exclusion Criteria:

* Simultaneous participation in another clinical study or participation in another clinical study before inclusion in the present study that could affect its objectives.
* Previous history of poor ovarian response (<4 oocytes retrieved) with a maximal dose of ovarian stimulation (≥300 IU/day).
* Use of hormone contraceptives in the month preceding eventual inclusion.
* Presence of a medical condition which is known to affect ART outcome (e.g. thyroid dysfunction).
* Active female smoking.
* Ongoing pregnancy.
* Current use of anti-depressants, anti-psychotics, steroids, antiepileptics or chemotherapy.
* Known allergy or hypersensitivity to any of the study non-IMP.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy women who have consented to a cycle of fresh oocyte donation and who have a total antral-follicle count (AFC) above 20 at the onset of ovarian stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Ocurrence of diferent features in the microtubule cytoskeleton | From October 2020 up to December 2020
  Both fresh and vitrified-warmed oocytes will be analysed in respect to: spindle morphology; chromosome congression at the metáfase plate; presence of microtubule aggregates and presence of pericentriolar material aggregates.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Nunes, PhD, Principal Investigator — Instituto Valenciano de Infertilidade de Lisboa
Locations (1):
- Instituto Valenciano de Infertilidade, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No